CLINICAL TRIAL: NCT02911207
Title: Evaluation of Emotion Management Skill Strengthening in Chronically Ill Patients, Benefiting From Creative and Physical Activities
Acronym: EvAd
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RC16_0011
Record Dates: First submitted 2016-08-25; First posted 2016-09-22 (Estimated); Last update posted 2021-06-21 (Actual); Status verified 2021-06

CONDITIONS: Emotion Management Skill; Educational Therapy; Creative and Physical Activities
Keywords: chronic ill patients; Emotion management skill; Quality of Life
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention arm (Experimental): patients choose one creative activity (evolutive art-therapy, writing workshop, theatre, singing) and one physical activity (pilates, mindfulness meditation, shiatsu, ayurvedic massage) that they will practice during the following six months
  Interventions: Behavioral: patients choose one creative activity and one physical activity
- control arm (Active Comparator): patients choose one creative activity (evolutive art-therapy, writing workshop, theatre, singing) and one physical activity (pilates, mindfulness meditation, shiatsu, ayurvedic massage) that they will practice during six months but they will start 6 months later after randomization
  Interventions: Behavioral: patients choose one creative activity and one physical activity

INTERVENTIONS:
Behavioral: patients choose one creative activity and one physical activity — taking part in 2 activities (a creative one and a physical one)

SUMMARY:
There are very few studies on emotion management in chronically ill patients. They usually include small sample size (less than 30 persons) and are not randomized controlled trials. However, emotion management is an essential coping skill in mental well-being and quality of life and is the subject of numerous studies in psychology.The investigators hypothesized that a creative and physical activities combination in chronically ill will promote the strengthening of emotion management skill. The investigators will conduct an innovating study combining quantitative and qualitative variables in a randomized controlled trial to confirm our hypothesis.

DETAILED DESCRIPTION:
1. Surveyors will conduct a first interview with patients (within an association "La Fabrique Créative de Santé" that provides free activities to chronically ill) , in order to collect data on emotion management and quality of life perception and to assess expectations regarding the activities. At the end of the interview, patients will be randomized in two groups.
2. In arm 1, patients choose one creative activity (evolutive art-therapy, writing workshop, theatre, singing) and one physical activity (pilates, mindfulness meditation, shiatsu, ayurvedic massage) that they will practice during the following six months.
3. In arm 2, patients will follow the same pattern but will start activities 6 months later.
4. After 6 months data on patients emotion management and quality of life perception will be collected again and interviews will be conducted regarding their overall satisfaction of the activities.
5. Every six months during one year, data will be collected by mail or e-mail.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old and over
* Chronical illness
* Followed by a physician from Nantes University hospital

Exclusion Criteria:

* Having already taken part in activities within the association "La Fabrique Créative de Santé"
* Mental illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2016-08-29 (Actual); Primary Completion 2018-12-04 (Actual); Study Completion 2018-12-04 (Actual)

PRIMARY OUTCOMES:
DERS questionnaire | 6 months after baseline interview
  differences between initial and final answers (after 6 months of intervention) scale composed of 36 items in 6 dimensions

SECONDARY OUTCOMES:
Changes in quality of life: comparison between baseline assessment and assessment 2 | 6 months after baseline interview
  With following scale of quality of life: SeiQoL
Changes in quality of life: comparison between baseline assessment and assessment 2 | 6 months after baseline interview
  With following scale of quality of life: EQ5D
Changes in quality of life: comparison between baseline assessment and assessment 2 | 6 months after baseline interview
  With following scale of quality of life: WHOQoL

CONTACTS AND LOCATIONS:
Locations (1):
- Nantes University Hospital, Nantes, Loire-Atlantique, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Le Rhun A, Caillet P, Lebeaupin M, Duval M, Guilmault L, Anthoine E, Borghi G, Leclere B, Moret L. Mind-body and art therapies impact on emotional regulation in patients with chronic diseases: a pragmatic mixed-methods randomized controlled trial. BMC Complement Med Ther. 2023 Sep 28;23(1):344. doi: 10.1186/s12906-023-04173-8. PMID 37770881